CLINICAL TRIAL: NCT05911789
Title: A Prospective Study to Evaluate Online Adaptive Radiotherapy in Rectal Cancer
Brief Title: Online Adaptive Radiation Therapy for Rectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-rectal cancer
Record Dates: First submitted 2023-05-25; First posted 2023-06-22 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; adaptive radiation therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online adaptive radiation therapy (Experimental): Patients receive adaptive radiotherapy therapy and concurrent chemotherapy.
  Interventions: Radiation: Online adaptive radiation therapy

INTERVENTIONS:
Radiation: Online adaptive radiation therapy — A dose of 45Gy will be delivered to planning target volume (PTV)
  Other Names: ART

SUMMARY:
In the present study, the investigators will evaluate the efficacy, toxicities, and of online adaptive radiation therapy (ART) for patients with rectal cancer treated with neoadjuvant chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. Diagnose with rectal cancer;
3. T3-T4 or N+, and no distant metastasis
4. Neoadjuvant chemoradiotherapy intended;
5. Surgery is expected after neoadjuvant therapy;
6. ECOG score 0-2, expected to lie in the treatment bed for at least half an hour;

Exclusion Criteria:

1. With contraindications to rectal MRI;
2. Received surgery, radiotherapy or chemotherapy for rectal cancer;
3. History of pelvic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-05 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities(CTCA | 3 months for the start of treatment
  evaluated with Common Terminology Criteria for Adverse Events (CTCAE) 5.0
Response rate after surgery | 3 monsh after treatment
  Clinical and pathological complete response and partial response rate after chemoradiotherapy

SECONDARY OUTCOMES:
Chronic toxicity | 2 years after treatment
  evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme
Dose coverage of target volume (assessed by planing target volume V100%) | Through study completion, an average of five month
  Planing target volume V100%, defined as the planing target volume receiving at least 100% of the prescribed dose (V100%), is used to evaluate the dose coverage of target volume.
Margins for clinical target volume(CTV) and gross tumor volume (GTV) | Through study completion, an average of five month
  Margins needed in online ART for CTV to planning clinical target volume (PCTV) and GTV to planning gross tumor volume (PGTV) to cover inter/intra-fraction motion

IPD SHARING:
Plan to Share IPD: Undecided